CLINICAL TRIAL: NCT04602208
Title: FOCAL HIGH-INTENSITY FOCUSED ULTRASOUND FOR PRIMARY LOCALIZED PROSTATE CANCER: MIDTERM ONCOLOGICAL OUTCOMES
Acronym: Focal HIFU for
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0960
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focal HIFU for primary localized prostate cancer: Between November 2009 and December 2016, at Edouard Herriot Hospital (Lyon, France), 146 consecutive patients were treated with focal HIFU for primary localized prostate cancer. Focal therapy was offered for low or intermediate risk disease (inclusion criteria: one tumor localized by systematic and targeted biopsies based on MRI findings, Gleason ≤7). Treatment failure was defined as local or systemic salvage treatment, a positive biopsy Gleason score of 7 or greater in-field or out-of-field in nontreated patients, prostate cancer metastasis or prostate cancer specific death.
  Interventions: Procedure: Retrospectively review of medical data in patients treated by focal HIFU for primary localized prostate cancer

INTERVENTIONS:
Procedure: Retrospectively review of medical data in patients treated by focal HIFU for primary localized prostate cancer — This study concern the patients with localized prostate cancer treated by Focal HIFU for low or intermediate risk disease. Three surgeons experienced in HIFU performed the procedures. Patients were treated with the Ablatherm device [EDAP TMS S.A., Vaulx-en-Velin, France] until July 2013 and then with the Focal-One device [EDAP TMS S.A.]. The data of all the patients treated between November 2009 to December 2016, at Edouard Herriot Hospital (Lyon, France), were prospectively maintain within a central database and retrospectively reviewed. The study primary outcome was retreatment-free survival (RFS) defined as any additional further treatment: local (FT/PGA for in-field or out-of-field recurrences or radical prostatectomy or external beam radiotherapy or whole gland HIFU) or systemic salvage treatment, a positive biopsy revealing PCa with an ISUP grade≥ 2 in nontreated patients, PCa metastasis or PCa specific death. The adverse events and functional outcomes were also evaluated.

SUMMARY:
Single-center evaluation of all patients treated for primary localized prostate cancer with focal HIFU from November 2009 to December 2016. To evaluate midterm oncological outcomes of focal HIFU therapy in low an intermediate risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* • The patients with low or intermediate risk PCa (PSA <20 ng/ml, Gleason score 7 or less and clinical stage T2b or less) who received PGA/FT using HIFU were included.

Exclusion Criteria:

* Patients who were previously treated with radiotherapy, androgen deprivation therapy (ADT) or other treatment for their prostate cancer were excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with low or intermediate risk PCa (PSA <20 ng/ml, Gleason Score 7 or less and clinical stage T2b or less) who received PGA/FT using HIFU
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Retreatment-free survival (RFS) | May 1, 2020
  The study primary outcome was retreatment-free survival (RFS) defined as any additional further treatment: local (FT/PGA for in-field or out-of-field recurrences or radical prostatectomy or external beam radiotherapy or whole gland HIFU) or systemic salvage treatment, a positive biopsy revealing PCa with an ISUP grade≥ 2 in nontreated patients, PCa metastasis or PCa specific death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France